CLINICAL TRIAL: NCT00740025
Title: A Prospective Randomized Study of QD vs BID Dosing in ART
Brief Title: Once Daily vs Twice Daily Administration of Gonadotropins in Assisted Reproductive Technologies (ART)
Acronym: QD vs BID
Status: Completed | Type: Observational
Sponsor: Virginia Center for Reproductive Medicine (Other)
Responsible Party: Fady I. Sharara, Virginia Center for Reproductive Medicine
Other Study IDs: 1-Sharara
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Pregnancy
Keywords: QD dose; BID dosing; peak estradiol; oocytes; implantation rate; pregnancy rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- QD: Women who received their meds as QD administration
- BID: Women who received their gonadotropins as a BID dose

SUMMARY:
This is a prospective randomized study evaluating dosing frequency of gonadotropin administration in ART cycles.

DETAILED DESCRIPTION:
Using once daily or bid dosing of gonadotropins in ART has been arbitrary with no studies showing whether splitting the medication dose improves ART parameters. This study was undertaken to provide an answer to this important question.

ELIGIBILITY:
Inclusion Criteria:

* women < 40 undergoing ART

Exclusion Criteria:

* women > 40
* endometriomas
* severe cervical stenosis
* testicular sperm

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between 21-40 yo
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 1 year

SECONDARY OUTCOMES:
peak estradiol, number of follicles, number of oocytes, implantation rate, multiple pregnancy rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fady I Sharara, M.D, Principal Investigator — Virginia Center for Reproductive Medicine
Locations (1):
- Virginia Center for Reproductive Medicine, Reston, Virginia, United States